CLINICAL TRIAL: NCT02808611
Title: Konditionerende Smertestimuli - Sammenligning af Forskellige Test og Konditioneringsmodaliteter
Brief Title: Influence of Propranolol on Conditioned Pain Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristian Kjær Petersen (Other)
Responsible Party: Sponsor-Investigator, Kristian Kjær Petersen, M.Sc, Ph.d., Aalborg University
Organization: Aalborg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: N-20150055
Record Dates: First submitted 2016-06-15; First posted 2016-06-22 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol (Active Comparator): Propranolol is a beta-blocker
  Interventions: Drug: propranolol
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: propranolol — Reduction of the ANS response
  Arms: Propranolol
Drug: Placebo
  Arms: Placebo

SUMMARY:
An extensive amount of studies indicate that conditioned pain modulation (CPM) test paradigms can be of use to evaluate the efficacy of the endogenous pain inhibition pathway in healthy controls and pain patients. A number of studies indicate that the autonomic nervous system (ANS) responds to painful stimulation by parasympathetic activity withdrawal and up-regulation of sympathetic activity (flight-or-fight mode), but it remains unknown whether these responses predict individual pain susceptibility or CPM efficacy and whether different pain modalities evoke different physiological stress responses, i.e. do individuals with low pain tolerance exhibit more vigorous ANS responses when subjected to controlled acute pain stimuli, and do high ANS responsiveness to pain coincide with altered psychophysical pain levels/CPM efficacy.

This study aims to investigate the effect of ANS responsiveness on CPM paradigms and to investigate if an exogenous, pharmaceutically induced decrease in the sympathetic drive of the ANS will yield decreased CPM efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous history of neurologic, musculoskeletal, mental illnesses or a chronic pain condition
* Lack of ability to cooperate
* Current use of medications that may affect the trial, e.g., analgesics, anti-inflammatory drugs
* Consumption of alcohol, caffeine, nicotine or painkillers the morning and until termination of the study on the study day
* Recent history of acute pain affecting the lower limb
* Participation in other pain trials throughout the study period
* Known diagnosis of cardio vascular diseases (low blood pressure, heart conditions)
* Asthma
* Decreased function of liver and kidneys
* Diabetes

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
CPM efficacy | 1-2 hours after propranolol/placebo and after 10 minutes break.
  A test stimuli will be applied and compared with a test stimuli simultaneous a condition stimuli.

SECONDARY OUTCOMES:
Temporal summation of pain | 1-2 hours after propranolol/placebo and after 10 minutes break.
  10 stimuli will be applied and subjects will back asked to rate the pain for each individual stimuli.
Heart-rate variability | 1-2 hours after propranolol/placebo and after 10 minutes break.
  Two-point Heart-rate variability recording will be conducted using the Polar RS800CX heart rate monitor.
Offset analgesia | 1-2 hours after propranolol/placebo and after 10 minutes break.
  Temperatures ranging from 45-48°C will be applied to the forearm in three phases (phase 1: 5 seconds, phase 2: 5 seconds, and phase 3: 20 seconds). The subjects will be asked to assess the pain of the thermal stimuli using the electronic VAS scale.

CONTACTS AND LOCATIONS:
Overall Officials: KRISTIAN K PETERSEN, Ph.D., Principal Investigator — Aalborg University
Locations (1):
- Center for Sensory Motor Interaction, Aalborg University, Aalborg East, Denmark

REFERENCES:
- [Derived] Petersen KK, Andersen HH, Tsukamoto M, Tracy L, Koenig J, Arendt-Nielsen L. The effects of propranolol on heart rate variability and quantitative, mechanistic, pain profiling: a randomized placebo-controlled crossover study. Scand J Pain. 2018 Jul 26;18(3):479-489. doi: 10.1515/sjpain-2018-0054. PMID 29858911